CLINICAL TRIAL: NCT03375892
Title: A Phase II Study of the Use of Deep Inspiration Breath Hold and Prone Irradiation to Decrease Cardiac Radiation Exposure
Brief Title: The Use of Deep Inspiration Breath Hold and Prone Irradiation to Decrease Cardiac Radiation Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Adam Currey, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00030436
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ; Invasive Breast Cancer
Keywords: radiation; Deep Inspiration Breath Hold; stage I; stage II; stage IIa
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prone Position with DIBH (Active Comparator): For prone positioning, patients will be positioned with alpha cradle casts, and a prone breast board.
  Interventions: Other: Deep Inspiration Breath Hold during Radiation
- Supine Position with DIBH (Active Comparator): For the supine positioning, patients will be positioned with the breast board currently in use in the Department of Radiation Oncology.
  Interventions: Other: Deep Inspiration Breath Hold during Radiation
- Prone Position with no DIBH (Active Comparator): For prone positioning, patients will be positioned with alpha cradle casts, and a prone breast board.
  Interventions: Other: Free breathing during radiation
- Supine Position with no DIBH (Active Comparator): For the supine positioning, patients will be positioned with the breast board currently in use in the Department of Radiation Oncology.
  Interventions: Other: Free breathing during radiation

INTERVENTIONS:
Other: Deep Inspiration Breath Hold during Radiation — The DIBH technique involves the patient breathing to a specified threshold and then holding that level of inspiration during every radiation therapy field delivered.
  Arms: Prone Position with DIBH; Supine Position with DIBH
Other: Free breathing during radiation — The patient will be instructed to breathe freely.
  Arms: Prone Position with no DIBH; Supine Position with no DIBH

SUMMARY:
This study aims to discover more about radiation techniques for people treated for left-sided breast cancer that minimizes exposure to the heart, as noted by mean heart dose.

DETAILED DESCRIPTION:
This study aims to discover more about radiation techniques for people treated for left-sided breast cancer that minimizes exposure to the heart, as noted by mean heart dose. Both prone (lying face down) radiation and Deep Inspiration Breath Hold (DIBH) are more labor-intensive and usually require longer treatment times for patients than traditional supine (lying face up) free-breathing radiation treatments. Thus, identifying people that benefit most from these techniques can better utilize resources. This study compares supine and prone positioning, with or without DIBH, to further assess which positioning technique will achieve the lowest cardiac radiation doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically proven diagnosis of left-sided invasive breast cancer or ductal carcinoma in situ receiving breast/chestwall irradiation +/- regional nodal irradiation, or a right-sided invasive ductal cancer status post-mastectomy or lumpectomy who will be receiving breast/chest wall and nodal irradiation.
* Patients must have undergone breast conserving surgery (i.e. lumpectomy, partial mastectomy) or mastectomy prior to enrollment.
* Patients must be 18 years of age or older.
* Study entry must be prior to CT simulation.
* Per Medical College of Wisconsin Department of Radiation Oncology Standard of Care, women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable forms of contraception during radiation therapy. Patients under age 50 with a uterus and ovaries must have a negative serum pregnancy test within one week of planned CT simulation per Radiation Oncology Departmental guidelines prior to CT simulation.
* Patients must provide study specific informed consent prior to study entry.
* Patients must be able to hold their breath long enough to undergo CT simulation in DIBH (ten to fifteen seconds). The patient should also affirm they can lie in the prone position. This will be determined by the treating radiation oncologist, as per current standard of care.

Exclusion Criteria:

* Patients who are unable to hold their breath long enough to undergo CT simulation in DIBH. While this may affect patients with chronic obstructive pulmonary disease (COPD) and/or other respiratory conditions, the presence of these comorbidities alone will not exclude patients from enrollment so long as they can maintain breath hold long enough to perform DIBH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Changes in EKG parameters prior to, during or after radiation therapy. | Baseline, 6 weeks, 6 months and 12 months
  Changes in QRS wave form will be categorized as 'present' or 'absent' based on the presentation (or lack) of a r' wave, or notched r or s wave on the EKG tracing. QRS-T angle will be measured in degrees.

SECONDARY OUTCOMES:
Change in mitochondrial energy production, as measured in leukocytes (peripheral blood mononuclear cells) from patients prior to and after undergoing radiation therapy. | baseline, 6 weeks, and 6 and 12 months post-radiation therapy
  Mitochondrial energy production will be measured by determining oxygen consumption rate (pmol of O2 consumed per second per·10^6 cells).
Changes in left ventricular ejection fraction prior to, during or after radiation therapy. | Baseline and 12 months
  This will be measured as a percentage.
Changes in left atrial volume prior to, during or after radiation therapy. | Baseline and 12 months
  This will be measured in millimeters.
Left ventricular wall thickness prior to, during or after radiation therapy. | Baseline and 12 months
  This will be measured in millimeters.
Arterial and aortic stiffness. | Baseline and 12 months
  This will be assessed by measuring the ascending aortic diameters 3 cm above the aortic valve at end-diastole and end-systole in the 2D parasternal view.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Currey, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No